CLINICAL TRIAL: NCT06833775
Title: Evaluation of Neoadjuvant Therapy Efficacy and Postoperative Pathological Indicators in Esophageal Cancer Using CT and Multimodal MRI
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qujinrong, Clinical Professor, Henan Cancer Hospital
Other Study IDs: 2024-621
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the group of patients who achieved pathological complete response (pCR) following neoadjuvant
- the group of patients who did not achieve pCR following neoadjuvant therapy and surgery for esophage

SUMMARY:
This study aims to predict the efficacy of different types of neoadjuvant therapy and related postoperative pathological indicators in patients with esophageal cancer based on imaging parameters from CT and multimodal MRI, as well as clinical indicators collected before and after neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients with histopathological diagnosis of esophageal cancer.
2. Patients underwent neoadjuvant therapy before radical surgery for esophageal cancer: neoadjuvant chemotherapy, neoadjuvant chemoradiotherapy, neoadjuvant chemotherapy plus immunotherapy, neoadjuvant chemoradiotherapy plus immunotherapy.
3. All patients underwent CT and multimodal MRI examinations before and after neoadjuvant therapy.
4. The preoperative clinical data and postoperative pathological data are complete.

Exclusion Criteria:

1. Patients with other primary malignant tumors or previous anti-tumor treatment.
2. CT and MRI images with poor quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed with esophageal cancer by pathology at Zhengzhou University Affiliated Cancer Hospital from January 1, 2017 to December 31, 2024. Based on pre-treatment examinations such as endoscopic ultrasound, CT, MRI, and multidisciplinary consultation opinions, these patients underwent radical esophagectomy after receiving different kinds of neoadjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
CT and multimodal MRI in prediction of neoadjuvant therapy efficacy and postoperative pathological indicators in esophageal cancer | March 2025 - January 2030
  To evaluate the effectiveness of CT and multimodal MRI in determining the neoadjuvant therapy efficacy and postoperative pathological indicators in esophageal cancer.

IPD SHARING:
Plan to Share IPD: Undecided